CLINICAL TRIAL: NCT01127009
Title: A Phase I Study of Bortezomib in Combination With MEC (Mitoxantrone, Etoposide, and Intermediate-Dose Cytarabine) for Relapsed/ Refractory Acute Myelogenous Leukemia (AML)
Brief Title: Bortezomib, Mitoxantrone, Etoposide, and Cytarabine in Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE4909; NCI-2010-01203 (Other: National Cancer Institute); CASE4909 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Bortezomib; Mitoxantrone; Etoposide; Podophyllotoxin; Cytarabine; Flow Cytometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8 and 11; and mitoxantrone IV, etoposide IV over 1 hour, and intermediate-dose cytarabine IV over 6 hours on days 1-6. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Drug: mitoxantrone hydrochloride; Drug: etoposide; Drug: cytarabine; Other: flow cytometry

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; PS-341; VELCADE
Drug: mitoxantrone hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; dihydroxyanthracenedione; mitoxantrone HCl; Novantrone
Drug: etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; epipodophyllotoxin; VePesid; VP-16; VP-16-213
Drug: cytarabine — Given IV
  Other Names: ARA-C; ARA-cell; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: flow cytometry — Correlative studies

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as mitoxantrone, etoposide, and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with combination chemotherapy may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of bortezomib when given together with mitoxantrone, etoposide, and cytarabine in treating patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the DLT, MTD, and the recommended Phase 2 dose of bortezomib in combination with MEC in patients with relapsed/refractory AML.

SECONDARY OBJECTIVES:

I. To describe the non-dose limiting toxicities associated with bortezomib in combination with MEC in patients with relapsed/refractory AML.

II. To describe any preliminary evidence of clinical activity of this combination (CR rate) in relapsed/refractory AML.

III. To determine the median CD74 antigen expression in patients achieving a response versus those patients not achieving a response.

OUTLINE:

This is a dose-escalation study of bortezomib.

Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8 and 11; and mitoxantrone IV, etoposide IV over 1 hour, and intermediate-dose cytarabine IV over 6 hours on days 1-6. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4-5 weeks.

ELIGIBILITY:
Inclusion

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study; female subject is not lactating
* Male subject agrees to use an acceptable method for contraception for the duration of the study
* Relapsed or refractory AML (excluding acute promyelocytic leukemia), based on World Health Organization Classification; all other subtypes of AML will be eligible; refractory disease will be considered failure to respond to 2 cycles of induction chemotherapy (7+3 and 5+2); any number of relapses will be eligible
* No evidence of leptomeningeal disease; a lumbar puncture does not need to be performed unless there is clinical suspicion of leptomeningeal disease
* Previous treatment related toxicities must have resolved to Grade 1 (excluding alopecia)
* Liver enzymes (AST and ALT) can not be greater than 2.5 times the upper limits of normal (ULN), and total bilirubin =< 1.5 x ULN within 14 days of enrollment
* Renal function: Serum creatinine should be =< 1.5 x ULN within 14 days of enrollment
* No serious or poorly controlled medical conditions that could be exacerbated by treatment or that would seriously complicate compliance with the protocol
* ECOG performance status 0-3
* No peripheral neuropathy >= Grade 2 within 14 days of trial enrollment
* Echocardiogram or MUGAs scan demonstrating an ejection fraction >= 45%
* Patients with secondary AML, and patients with a prior autologous and allogeneic bone marrow transplant are eligible
* Patients with an allogeneic transplant must meet the following conditions: the transplant must have been performed more than 90 days before registration to this study, the patient must not have >= Grade 2 acute graft versus host disease (GvHD), or either moderate or severe limited chronic GvHD, or extensive chronic GvHD of any severity; the patient must be off all immunosuppression for at least 2 weeks
* No uncontrolled infections
* No history of hypersensitivity to boron or mannitol
* No known history of HIV or active hepatitis B or C
* No major surgery within 4 weeks prior to trial enrollment

Exclusion

* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant
* Patient has >= Grade 2 peripheral neuropathy within 14 days before enrollment
* Female subject is pregnant or breast-feeding; confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women
* Patient has received any standard or investigational therapy for their leukemia within 14 days before enrollment (except for hydrea)
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Patients with prior malignancy are eligible; however, the patient must be in remission from the prior malignancy and have completed all chemotherapy and radiotherapy at least 6 months prior to registration and all treatment-related toxicities must have resolved
* Leptomeningeal/ central nervous system involvement with AML; a lumbar puncture does not need to be performed unless there is clinical suspicion
* Patients who have had prior pulmonary radiation
* Prohibited Concurrent Therapy: any investigational agent other than VELCADE; G-CSF and GM-CSF are not allowed

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
MTD of bortezomib | two times a week until Day 28, then every week until Day 45 (+/- 2 days), then 4 wks after treatment.

SECONDARY OUTCOMES:
Non-dose limiting toxicities | two times a week until Day 28, then every week until Day 45 (+/- 2 days), then 4 wks after treatment.
CR/ CRp rate | repeated 4 weeks after the post-treatment bone marrow aspirate/biopsy.
CD74 antigen expression | to be performed only on the pre-treatment sample

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Advani, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States